CLINICAL TRIAL: NCT05481736
Title: Efficacy and Safety of COMP360 Psilocybin Therapy in Anorexia Nervosa: a Proof-of-concept Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: COMPASS Pathways (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMP 401
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 25 mg COMP360 Psilocybin (Experimental): 25 mg COMP360 Psilocybin
  Interventions: Drug: Psilocybin
- 1 mg COMP360 Psilocybin (Active Comparator): 1 mg COMP360 Psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — COMP360 Psilocybin administered under supportive conditions
  Other Names: COMP360

SUMMARY:
Efficacy and Safety of COMP360 Psilocybin therapy in Anorexia Nervosa: a Proof-of-concept Study

DETAILED DESCRIPTION:
This study aims to explore the efficacy and safety of COMP360 25 mg as compared to COMP360 1 mg (control condition) administered with psychological support in participants with Anorexia Nervosa

ELIGIBILITY:
Inclusion Criteria:

1. Any sex and aged 18 years or above at screening.
2. Meeting criteria for AN either restrictive or binge-purging type, according to the DSM-5, based on medical records, clinical assessment, BMI, and documented completion of MINI 7.0.2 and EDE at screening.
3. Have successfully discontinued all prohibited medications for a period of at least two weeks prior to baseline. For fluoxetine (Prozac), immediate cessation at screening period visit 1a followed by at least four weeks of washout will be required prior to baseline.
4. Has a history of disordered eating with duration of at least 3 years prior to screening, that is consistent with AN.
5. BMI ≥15 kg/m2 and ≤20 kg/m2. For participants with a BMI <16 kg/m2 and >18.5 kg/m2 at screening, approval from the Medical Monitor will be required. Any participant with a BMI >18.5 kg/m2 must meet all of the criteria for AN except that, despite significant weight loss, the individual's weight is within or above the normal range.
6. Being otherwise medically stable at screening determined by clinical interview, clinical laboratory values, vital signs, ECG, and medical history.
7. Have at least one documented prior attempt at treatment in the past 3 years.

Exclusion Criteria:

1. Prior or ongoing bipolar disorder, any psychotic disorder, including schizophrenia, schizophreniform disorder, schizoaffective disorder, brief psychotic disorder (unless substance induced or due to a medical condition), antisocial personality disorder, or any serious psychiatric comorbidity as assessed by medical history and a structured clinical interview (MINI 7.0.2).
2. Prior or ongoing paranoid, schizoid, schizotypal, histrionic, narcissistic personality disorder based on medical history and clinical judgment.
3. Borderline personality disorder as demonstrated by medical history, the MINI Plus - BPD and clinical judgment.
4. Significant suicide risk as defined by (1) suicidal ideation as endorsed on items 4 or 5 on the C-SSRS within the past year, at screening or at baseline, or; (2) suicidal behaviours within the past year or; (3) clinical assessment of significant suicidal risk during participant interview.
5. Current (within last year) alcohol or substance use disorder as informed by the DSM-5 assessed via the MINI 7.0.2, and urine toxicology at screening.
6. Other personal circumstances and behaviour judged to be incompatible with establishment of rapport or safe exposure to psilocybin.
7. Exposure to psilocybin, or any other psychedelics, such as ayahuasca, mescaline, LSD, or peyote within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Eating Disorder Examination (EDE) global score | Week 4
  The EDE is a structured clinical interview (investigator rated) used to measure severity of the characteristic psychopathology of eating disorders

SECONDARY OUTCOMES:
Safety | Up to 12 weeks
  Proportion of patients with adverse events (AEs)
Change from baseline in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Week 4
  The Y-BOCS self-rated version consists of a 10 item measure with a total score ranging from 0 to 40, with higher scores indicating increased severity of symptoms
Change from baseline in weight | Up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Altman Clinical and Translational Research Institute, San Diego, California
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Dell Medical School, Austin, Texas
- Tallaght University Hospital, Dublin, Ireland
- Kings College London, Institute of Psychiatry, Psychology and Neurology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided